CLINICAL TRIAL: NCT05691608
Title: MoleculAr Profiling for Pediatric and Young Adult Cancer Treatment Stratification 2
Acronym: MAPPYACTS2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A02990-41; 2021-3321 (Other: CSET NUMBER)
Record Dates: First submitted 2022-12-12; First posted 2023-01-20 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor; Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with solid tumor or leukemia (no treatment) (Experimental): Patient with solid tumor or leukemia (no treatment)
  Interventions: Biological: Solid tumor and CT DNA

INTERVENTIONS:
Biological: Solid tumor and CT DNA — Biopsy and blood sample

SUMMARY:
FMG2025 continues the previous efforts to propose treatment for patients based on the molecular characteristics of their tumor at treatment failure in cancer precision medicine trials within standard of care in France. However, whereas FMG2025 is a descriptive effort providing the basis for clinical decisions, MAPPYACTS 2 will translate these findings to clinical actions. The symbiosis is critical to advance patient care.

Since 2012, the molecular profiling trials "MOlecular Screening for CAncer Treatment Optimization" (MOSCATO-01) and "MoleculAr Profiling for Pediatric and Young Adult Cancer Treatment Stratification" (MAPPYACTS) have included pediatric and adolescent patients with recurrent or refractory malignancy that underwent on-purpose biopsy or surgical intervention. Whole Exome Sequencing of tumor and normal tissue and RNA Sequencing of tumor tissue have been applied to detect genomic alterations that could lead to an adapted targeted treatment. Furthermore, ancillary studies were associated exploring circulating tumor DNA, the immune contexture of tumors and developing Patient-Derived Xenografts (PDX).

The FMG2025 project transfers the molecular profiling of advanced pediatric cancers into a global approach that is now considered standard of care in France. Subsequent clinical recommendations and decisions will be made based on discussions with biologists, scientist and physicians in the molecular and clinical molecular tumor boards. Associated ancillary research studies and links to clinical interventional studies remain essential elements of the program to provide clinical, translational and basic research in order to improve scientific knowledge.

The program is articulated in two main parts that are closely interacting:

FMG2025 - Cancers et leucémies pédiatriques en échec de traitement or equivalent international projects that cover the sequencing of tumor and blood samples and provide molecular reports.

The clinical study MAPPYACTS 2 that provides clinical and therapeutic discussions of the sequencing results and therapy recommendations via the clinical molecular tumor board reports. It collects molecular and comprehensive clinical data of the patients registered in FMG2025 or equivalent international projects and thereby constitutes the critical link to clinical interventional studies and its sponsors ensuring facilitated access to these trials. It also covers and coordinates ancillary research studies.

DETAILED DESCRIPTION:
MAPPYACTS 2 is a prospective international multicentric clinical study to provide clinical therapeutic recommendations, to set up the molecular and comprehensive clinical database of patients with relapsed or refractory pediatric malignancies in FMG2025 - Cancers et leucémies pédiatriques en échec de traitement or equivalent international projects, to collect the follow-up data on treatment and patients' outcome, in order to determine the outcome of the program in regard to benefit to the patient, all the patients and to health care. It will also serve as a central link to interventional study platforms and international precision medicine programs, and to cover and coordinate ancillary research studies that lead to improved treatment and outcome for children with advanced malignancies.

Subsequent clinical recommendations and decisions will be made based on discussions with biologists, scientists and physicians in the molecular and clinical molecular tumor boards run by the MAPPYACTS 2 study teams.

Associated ancillary research studies and links to clinical interventional studies are essential components of the program to perform clinical, translational and basic research in order to generate scientific knowledge and develop new treatment strategies that improve outcome of these patients. Research projects will be discussed and agreed on in the MAPPYACTS 2 study committee.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for sequencing of the tumor within the FMG2025 or equivalent program and written informed consent for FMG2025 "Cancers et leucémies pédiatriques en échec de traitement" or equivalent, according to local regulations
* Written informed consent of MAPPYACTS 2 to collect molecular and comprehensive clinical data on cancer diagnosis, therapies, therapy outcomes, to provide clinical therapeutic recommendations, to collect follow-up data on treatment and patients' outcome; optional written consents to perform to ancillary research studies, according to local regulations. The written consent will include access to reimbursement data from the French national health insurance through linkage with the Système National des Données de Santé (SNDS) or equivalent.
* Patient with histologically/cytologically confirmed solid tumor or leukemia which is relapsed or refractory to standard treatment and who is potentially eligible for an experimental treatment or an early phase clinical trial
* Planned tumor biopsy, surgical resection, bone marrow or blood sample or recently (preferably within the last 3 months) archived frozen tumor material available of the current recurrent or refractory disease
* Patients aged ≤ 25 years at the time of initial diagnosis
* Performance status and life expectancy > 3 months expected to allow enrolment into an clinical trial
* Patients affiliated with a Social Security Regimen or beneficiary of the same, as per local regulatory requirements

Exclusion Criteria:

* Any concurrent illness or laboratory abnormality that, in the opinion of the investigator, is likely to interfere with the interpretation of study results
* Pregnant women

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1800 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2030-09-09 (Estimated); Study Completion 2030-09-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 3 years
  Defined as the time from study entry to death whatever the cause of death, after 3 years, for the whole cohort and according to cancer type.
The number of additional technologies and new treatment strategies that are introduced in the care for advanced pediatric cancers through this research program. | 3 years
  The number of patients receiving matched targeted treatments The number of new treatment strategies that are introduced in the care for advanced pediatric cancers through this research program The number of additional technologies that are introduced in the care for advanced pediatric cancers through this research program
The types of additional technologies and new treatment strategies that are introduced in the care for advanced pediatric cancers through this research program. | 3 years
  The type of patients receiving matched targeted treatments The type of new treatment strategies that are introduced in the care for advanced pediatric cancers through this research program The type of additional technologies that are introduced in the care for advanced pediatric cancers through this research program

SECONDARY OUTCOMES:
Objective response rate on treatment attributed by the molecular tumor board in the clinical trial, overall and according to the treatment decision | 3 years
  Objective tumor response measured according to the standard for each tumor entity (i.e. RECIST 1.1, INRC, RANO, etc.).
  Assessed for the whole cohort, for each disease entity as well as for each suggested treatment and until last follow-up.
  The number and proportion of patients that are suggested to receive a matched targeted agent Direct medical costs including the planned or recently performed intervention
Progression-free survival (PFS) | 3 years
  Defined as the time interval from start of attributed treatment (targeted or not) to progression or death.
  They will be assessed for the whole cohort, for each disease entity as well as for each suggested treatment and until last follow-up.
5-year overall survival | 5 years
  Defined as the time from study entry to death whatever the cause of death, after 5 years.
  They will be assessed for the whole cohort, for each disease entity as well as for each suggested treatment and until last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit GEOERGER, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (29):
- France (29):
  - Gustave Roussy, Paris, Villejuif
  - CHU Amiens-Picardie, Amiens
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CHU Pellegrin, Bordeaux
  - CHRU Morvan, Brest
  - CHU de Caen, Caen
  - CHU Estaing, Clermont-Ferrand
  - CHU Dijon François Mitterand, Dijon
  - CHU Grenoble Alpes, Grenoble
  - Centre Oscar Lambret, Lille
  - Chu Limoges, Limoges
  - IHOP, Lyon
  - CHU La Timone, Marseille
  - CHU Arnaud de Villeneuve, Montpellier
  - CHU Nantes, Nantes
  - CHU de Nice, Nice
  - Institut Curie, Paris
  - Hopital Armand Trousseau, Paris
  - CHU Poitiers, Poitiers
  - CHU Reims- Hôpital Américain, Reims
  - CHU Rennes Hôpital Sud, Rennes
  - CHU de Rouen, Rouen
  - CHU de La Réunion site nord, Saint-Denis
  - CHU Saint Etienne, Saint-Etienne
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital des Enfants - CHU de Toulouse, Toulouse
  - Hôpital Clocheville, Tours
  - CHRU Nancy Hôpital Enfants, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Study protocol Informed Consent Form
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available in January 2023 The duration of the availability is up to 2030.